CLINICAL TRIAL: NCT00328393
Title: Effect of Pioglitazone on Ambulatory Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-000570-52
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension; Diabetes Mellitus Type 2
Keywords: Hypertension
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Pioglitazone (Active Comparator): Pioglitazone 45 mg, 8 weeks
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 45 mg 8 weeks
  Arms: Pioglitazone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The anti-diabetic pioglitazone has been found to reduce casual blood pressure. To date, no data are available looking at this effect in detail. Especially, ambulatory blood pressure has not yet been utilized to confirm the hypothesis that pioglitazone has blood pressure lowering effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 years
* Diabetes mellitus Type 2 (HbA1c 7 - 8.5%)
* Casual blood pressure > = 130/80 mmHg, < 160/100 mmHg

Exclusion Criteria:

* Therapy with insulin
* Combination therapy of sulfonyl-urea und metformin
* Therapy with nateglinid, repaglinid or an other substance of this drug family
* Allergy against pioglitazone or other composites of the tablet
* History of heart failure (NYHA I bis IV)
* Hepatic insufficiency
* Transaminases > 2.5-fold of the upper normal limit
* End-stage renal failure
* Syndrome of polycystic ovaries
* Absence of effective contraception in women of childbearing potential
* Pregnancy or breast-feeding

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-03; Primary Completion 2007-03 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Median of systolic 24-hour ambulatory blood pressure | 8 weeks
  Change of 24-hour blood pressure after 8 weeks of treatment

SECONDARY OUTCOMES:
Median of 24-hour diastolic ambulatory blood pressure | 8 weeks
  Change of 24-hour diastolic blood pressure after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, Prof., Principal Investigator — University of Erlangen-Nürnberg, Medical Department 4
Locations (1):
- CRC Medical Department IV, Erlangen, Germany